CLINICAL TRIAL: NCT06630650
Title: A Single Center Prospective Natural History and Outcome Measure Validation Study of Congenital Myasthenic Syndromes
Brief Title: A Prospective Natural History and Outcome Measure Validation Study of Congenital Myasthenic Syndromes
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10002093; 002093-N
Record Dates: First submitted 2024-10-06; First posted 2024-10-08 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10-17

CONDITIONS: Myasthenic Syndromes, Congenital
Keywords: Congenital Myasthenic Syndrome; Collagen Q; Downstream of tyrosine kinase 7; DOK7; COLQ
MeSH Terms: conditions — Myasthenic Syndromes, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COLQ-related CMS: Genetically confirmed COLQ-related CMS

SUMMARY:
Background:

Congenital myasthenic syndromes (CMSs) are a group of inherited disorders that affect how the nerves communicate with muscles. These can cause many problems that affect how people can move and use their bodies.

Objective:

This is a natural history study to learn more about how CMSs affect the body and cause changes over time.

Eligibility:

People aged 6 months or older with a CMS. The study will focus on DOK7- and COLQ-related CMSs, as well as other forms.

Design:

Participants will have up to 7 visits in 5 years. At each visit, participants will undergo many tests, including:

Physical exam with blood and urine tests.

Tests of their heart and lung function.

Exams of the eyes, lungs, muscles, and nerves. These will be done with different specialists.

Exams of the arms and hands and of body use and movements. These will also be done with specialists.

Photos and videos may be taken.

Muscle ultrasound. Participants will lie still as a wand is rubbed over their skin.

Magnetic resonance imaging (MRI) scans. Participants will lie still on a bed that slides partway into a large tube. A parent or other person may remain in the room, too. The scan will take 60 minutes.

Electromyography (EMG). Participants will lie still or may be asked to move around. A machine will measure the electrical activity in their muscles.

An activity monitor may be placed on the participant s wrist, ankle, or hip for up to 2 weeks. The monitor is about the size of a wristwatch.

A sample of skin may be removed....

DETAILED DESCRIPTION:
Study Description:

This natural history and outcome measure validation study aims to longitudinally characterize the clinical manifestations of all congenital myasthenic syndromes (CMS), with a focus on DOK7 and COLQ-related CMS. Both are ultra-rare inherited disorders of the neuromuscular junction. This study will also assess the validity and interrater reliability of outcome measures to support clinical trial readiness in these populations.

Primary Objective:

Characterize baseline clinical manifestations and CMS disease course over one year.

Co-Primary Objective:

Assess the validity and interrater reliability of outcome measures in CMS.

Secondary Objectives:

Characterize the extended disease course of CMS (Years 2 through 5)

Exploratory Objectives:

Biomarker identification, accelerometer validation, and MCID estimation.

Primary Endpoints:

Change from baseline to Year 1 in the following (as age-appropriate and tolerated-performed in all participants unless age ranges specified):

* Physical strength

  * MRC scale (all; as tolerated/developmentally appropriate)
  * Quantitative muscle assessment of shoulder abductors, elbow flexors/extensors, hip flexors and knee extensors/flexors (QMA >=7y)
  * Myotools grip and pinch strength (>=6y)
* Physical performance

  * Six-minute walk test distance (>=6y)
  * Repeated 1 minute sit to stand (>=2y)
  * Performance of Upper Limb (PUL) (>=2y)
  * Time of outstretched arm (>=2y)
* Disease severity

  --Quantitative Myasthenia Gravis (QMG) Score (>= 12y)
* Motor function <2y

  * Hammersmith infant neurological scale score (<2y)
  * Sitting balance score (<2y)
* Motor function >2y

  * Motor function measure score (MFM20, 2-6y) (MFM32, >=7y)
  * Time to ascend four stairs, descend four stairs, supine to stand (>=5y)
* Development

  --Developmental motor scale quotients (<5y)
* Pulmonary function >=5y

  * Forced vital capacity (FVC)
  * Slow vital capacity (SVC)
  * Forced vital capacity at 1 second (FEV1)
  * Maximum inspiratory and expiratory pressures (MIP/MEP)
  * End-tidal CO2 (ETCO2)
* Quality of life

  * Myasthenia Quality of Life (PM-QOL15 <18y, MG-QOL15 >=18)
  * PROMIS-57 Profile (>=18y)
  * PROMIS Ped-25 Profile (8-17y)
  * PROMIS Parent Proxy CAT (5-7y)
  * NeuroQoL (fatigue and upper and lower limb function domains, (>=8y)
  * MG-ADL (>=18y)
* Serious adverse and disease-related events

  * Narrative clinician description
  * Causality assessment (related or unrelated to the research or disease)
  * Event severity (CTCAE v5)
  * Event MedDRA system organ class, and preferred term

Co-Primary Endpoints:

Interrater reliability in physical strength, physical performance, motor function, and quality of life primary endpoints.

Secondary Endpoints:

Change over time in primary endpoints (Years 2 through 5).

Exploratory Endpoints:

* Physical performance

  * Timed up and go (TUG) test x3 (>=2y)
  * Wearable sensor metrics during physical performance tests
* Biomechanics

  * Stride length, cadence, velocity captured in clinic by wearable device
  * Stride velocity 95th centile
* Free-living physical activity

  * Endpoints collected over 2-week data capture period will include:
  * Number of sit-to-stand transitions
  * Step count
  * Average cadence per walking episode
  * Number of falls
  * Activity counts (light, moderate, vigorous, moderate to vigorous)
  * Upper limb movements
  * Proposal to use in infants/toddlers, use of one device/chest strap.
* Ophthalmology

  * Marginal reflex distance (Ptosis)
  * Pupillometry
  * Ocular Motility utilizing Modified Goldmann Perimeter per NEI
* Quality of life

  * CMS-ST- Infant/Young Child 6 months - <=3 years of age
  * CMS-ST Child/Adult (4 years - <=18 years)
* Biomarkers

  * Peripheral biomarkers
  * Optional skin punch biopsy (fibroblast culture)
* Imaging

  * Muscle MRI lower extremities (T1 and Dixon)
  * Muscle ultrasound (echogenicity)
* Nerve function

  --EMG/NCS (sfEMG and RNS)
* Measurement of AE burden

  * Adverse Event Unit (AEU)

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged >= 6 months of age
* Clinically stable as evidenced by medical record review and remote screening questionnaire
* Genetically confirmed congenital myasthenic syndrome (pathogenic or likely pathogenic variants identified by CLIA testing in an established CMS-related gene including but not limited to DOK7, COLQ, CHRNE, RAPSN, CHAT, GFPT1, DPAGT1 OR pathogenic/likely pathogenic variant in combination with a variant of uncertain significance (VUS) AND additional clinical supporting evidence of CMS).
* Agreement to adhere to Lifestyle Considerations throughout study duration
* Ability of subject to understand and the willingness to provide informed consent (>=18 years of age) and assent (>=7 years of age).

EXCLUSION CRITERIA:

* Received gene transfer therapy
* Pregnant women (prior to enrollment)
* Ongoing medical condition or medication use that is deemed by the Principal Investigator to interfere with the conduct or assessments of the study or safety of the subject.

Ages: 6 Months to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with congenital myasthenic syndromes with a focus on DOK7 and COLQ subtypes.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2042-12-02 (Estimated); Study Completion 2044-12-02 (Estimated)

PRIMARY OUTCOMES:
Characterize baseline clinical manifestations and CMS disease | One year
Assess the validity and interrater reliability of outcome measures in CMS | 5 Years

SECONDARY OUTCOMES:
Characterize the extended disease course of CMS | Years 2-5

CONTACTS AND LOCATIONS:
Overall Officials: Carsten G Bonnemann, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brooks PJ, Ottinger EA, Portero D, Lomash RM, Alimardanov A, Terse P, Xu X, Chandler RJ, Geist Hauserman J, Esposito E, Bonnemann CG, Venditti CP, Austin CP, Pariser A, Lo DC. The Platform Vector Gene Therapies Project: Increasing the Efficiency of Adeno-Associated Virus Gene Therapy Clinical Trial Startup. Hum Gene Ther. 2020 Oct;31(19-20):1034-1042. doi: 10.1089/hum.2020.259. No abstract available. PMID 32993373
- [Background] Nicole S, Azuma Y, Bauche S, Eymard B, Lochmuller H, Slater C. Congenital Myasthenic Syndromes or Inherited Disorders of Neuromuscular Transmission: Recent Discoveries and Open Questions. J Neuromuscul Dis. 2017;4(4):269-284. doi: 10.3233/JND-170257. PMID 29125502
- [Background] Maggi L, Bernasconi P, D'Amico A, Brugnoni R, Fiorillo C, Garibaldi M, Astrea G, Bruno C, Santorelli FM, Liguori R, Antonini G, Evoli A, Bertini E, Rodolico C, Mantegazza R. Italian recommendations for diagnosis and management of congenital myasthenic syndromes. Neurol Sci. 2019 Mar;40(3):457-468. doi: 10.1007/s10072-018-3682-x. Epub 2018 Dec 15. PMID 30554356
- [Background] Bergamin E, Hallock PT, Burden SJ, Hubbard SR. The cytoplasmic adaptor protein Dok7 activates the receptor tyrosine kinase MuSK via dimerization. Mol Cell. 2010 Jul 9;39(1):100-9. doi: 10.1016/j.molcel.2010.06.007. PMID 20603078
- [Background] Sigoillot SM, Bourgeois F, Lambergeon M, Strochlic L, Legay C. ColQ controls postsynaptic differentiation at the neuromuscular junction. J Neurosci. 2010 Jan 6;30(1):13-23. doi: 10.1523/JNEUROSCI.4374-09.2010. PMID 20053883
- [Background] Hallock PT, Xu CF, Park TJ, Neubert TA, Curran T, Burden SJ. Dok-7 regulates neuromuscular synapse formation by recruiting Crk and Crk-L. Genes Dev. 2010 Nov 1;24(21):2451-61. doi: 10.1101/gad.1977710. PMID 21041412
- [Background] Palace J, Lashley D, Newsom-Davis J, Cossins J, Maxwell S, Kennett R, Jayawant S, Yamanashi Y, Beeson D. Clinical features of the DOK7 neuromuscular junction synaptopathy. Brain. 2007 Jun;130(Pt 6):1507-15. doi: 10.1093/brain/awm072. Epub 2007 Apr 23. PMID 17452375
- [Background] Lee M, Beeson D, Palace J. Therapeutic strategies for congenital myasthenic syndromes. Ann N Y Acad Sci. 2018 Jan;1412(1):129-136. doi: 10.1111/nyas.13538. PMID 29381222
- [Background] McMacken GM, Spendiff S, Whittaker RG, O'Connor E, Howarth RM, Boczonadi V, Horvath R, Slater CR, Lochmuller H. Salbutamol modifies the neuromuscular junction in a mouse model of ColQ myasthenic syndrome. Hum Mol Genet. 2019 Jul 15;28(14):2339-2351. doi: 10.1093/hmg/ddz059. PMID 31220253
- [Background] James MA. Use of the Medical Research Council muscle strength grading system in the upper extremity. J Hand Surg Am. 2007 Feb;32(2):154-6. doi: 10.1016/j.jhsa.2006.11.008. No abstract available. PMID 17275587
- [Background] Fernandez-Rhodes LE, Kokkinis AD, White MJ, Watts CA, Auh S, Jeffries NO, Shrader JA, Lehky TJ, Li L, Ryder JE, Levy EW, Solomon BI, Harris-Love MO, La Pean A, Schindler AB, Chen C, Di Prospero NA, Fischbeck KH. Efficacy and safety of dutasteride in patients with spinal and bulbar muscular atrophy: a randomised placebo-controlled trial. Lancet Neurol. 2011 Feb;10(2):140-7. doi: 10.1016/S1474-4422(10)70321-5. Epub 2011 Jan 6. PMID 21216197
- [Background] Bortolani S, Brusa C, Rolle E, Monforte M, De Arcangelis V, Ricci E, Mongini TE, Tasca G. Technology outcome measures in neuromuscular disorders: A systematic review. Eur J Neurol. 2022 Apr;29(4):1266-1278. doi: 10.1111/ene.15235. Epub 2022 Jan 10. PMID 34962693
- [Background] Bruggeman BS, Vincent HK, Chi X, Filipp SL, Mercado R, Modave F, Guo Y, Gurka MJ, Bernier A. Simple tests of cardiorespiratory fitness in a pediatric population. PLoS One. 2020 Sep 4;15(9):e0238863. doi: 10.1371/journal.pone.0238863. eCollection 2020. PMID 32886730
- [Background] Servais L, Mercuri E, Straub V, Guglieri M, Seferian AM, Scoto M, Leone D, Koenig E, Khan N, Dugar A, Wang X, Han B, Wang D, Muntoni F; SKIP-NMD Study Group. Long-Term Safety and Efficacy Data of Golodirsen in Ambulatory Patients with Duchenne Muscular Dystrophy Amenable to Exon 53 Skipping: A First-in-human, Multicenter, Two-Part, Open-Label, Phase 1/2 Trial. Nucleic Acid Ther. 2022 Feb;32(1):29-39. doi: 10.1089/nat.2021.0043. Epub 2021 Nov 17. PMID 34788571
- [Background] de Lattre C, Payan C, Vuillerot C, Rippert P, de Castro D, Berard C, Poirot I; MFM-20 Study Group. Motor function measure: validation of a short form for young children with neuromuscular diseases. Arch Phys Med Rehabil. 2013 Nov;94(11):2218-26. doi: 10.1016/j.apmr.2013.04.001. Epub 2013 Apr 18. PMID 23602884
- [Background] Berard C, Payan C, Hodgkinson I, Fermanian J; MFM Collaborative Study Group. A motor function measure for neuromuscular diseases. Construction and validation study. Neuromuscul Disord. 2005 Jul;15(7):463-70. doi: 10.1016/j.nmd.2005.03.004. PMID 16106528
- [Background] Tindall RS, Rollins JA, Phillips JT, Greenlee RG, Wells L, Belendiuk G. Preliminary results of a double-blind, randomized, placebo-controlled trial of cyclosporine in myasthenia gravis. N Engl J Med. 1987 Mar 19;316(12):719-24. doi: 10.1056/NEJM198703193161205. PMID 3547126
- [Background] Barohn RJ, McIntire D, Herbelin L, Wolfe GI, Nations S, Bryan WW. Reliability testing of the quantitative myasthenia gravis score. Ann N Y Acad Sci. 1998 May 13;841:769-72. doi: 10.1111/j.1749-6632.1998.tb11015.x. No abstract available. PMID 9668327
- [Background] Griffiths A, Toovey R, Morgan PE, Spittle AJ. Psychometric properties of gross motor assessment tools for children: a systematic review. BMJ Open. 2018 Oct 27;8(10):e021734. doi: 10.1136/bmjopen-2018-021734. PMID 30368446
- [Background] Richardson C, Smith T, Schaefer A, Turnbull D, Griffiths P. Ocular motility findings in chronic progressive external ophthalmoplegia. Eye (Lond). 2005 Mar;19(3):258-63. doi: 10.1038/sj.eye.6701488. PMID 15272295
- [Background] Chiang J, Mehta K, Amin R. Respiratory Diagnostic Tools in Neuromuscular Disease. Children (Basel). 2018 Jun 15;5(6):78. doi: 10.3390/children5060078. PMID 29914128
- [Background] Della Marina A, Wibbeler E, Abicht A, Kolbel H, Lochmuller H, Roos A, Schara U. Long Term Follow-Up on Pediatric Cases With Congenital Myasthenic Syndromes-A Retrospective Single Centre Cohort Study. Front Hum Neurosci. 2020 Dec 7;14:560860. doi: 10.3389/fnhum.2020.560860. eCollection 2020. PMID 33364925
- [Background] Prior DE, Cooper BA, Zhang B, Ghosh PS. Developing outcome measures of disease activity in pediatric myasthenia. Muscle Nerve. 2021 May;63(5):751-757. doi: 10.1002/mus.27208. Epub 2021 Feb 28. PMID 33604899
- [Background] Cella D, Choi SW, Condon DM, Schalet B, Hays RD, Rothrock NE, Yount S, Cook KF, Gershon RC, Amtmann D, DeWalt DA, Pilkonis PA, Stone AA, Weinfurt K, Reeve BB. PROMIS(R) Adult Health Profiles: Efficient Short-Form Measures of Seven Health Domains. Value Health. 2019 May;22(5):537-544. doi: 10.1016/j.jval.2019.02.004. PMID 31104731
- [Background] Cox ED, Connolly JR, Palta M, Rajamanickam VP, Flynn KE. Reliability and validity of PROMIS(R) pediatric family relationships short form in children 8-17 years of age with chronic disease. Qual Life Res. 2020 Jan;29(1):191-199. doi: 10.1007/s11136-019-02266-x. Epub 2019 Aug 10. PMID 31401748
- [Background] Varni JW, Thissen D, Stucky BD, Liu Y, Magnus B, Quinn H, Irwin DE, DeWitt EM, Lai JS, Amtmann D, Gross HE, DeWalt DA. PROMIS(R) Parent Proxy Report Scales for children ages 5-7 years: an item response theory analysis of differential item functioning across age groups. Qual Life Res. 2014 Feb;23(1):349-61. doi: 10.1007/s11136-013-0439-0. Epub 2013 Jun 6. PMID 23740167
- [Background] Finlayson S, Morrow JM, Rodriguez Cruz PM, Sinclair CD, Fischmann A, Thornton JS, Knight S, Norbury R, White M, Al-Hajjar M, Carboni N, Jayawant S, Robb SA, Yousry TA, Beeson D, Palace J. Muscle magnetic resonance imaging in congenital myasthenic syndromes. Muscle Nerve. 2016 Aug;54(2):211-9. doi: 10.1002/mus.25035. Epub 2016 Feb 22. PMID 26789134
- [Background] Ramdas S, Beeson D. Congenital myasthenic syndromes: where do we go from here? Neuromuscul Disord. 2021 Oct;31(10):943-954. doi: 10.1016/j.nmd.2021.07.400. PMID 34736634
- [Background] Benatar M, Sanders DB, Burns TM, Cutter GR, Guptill JT, Baggi F, Kaminski HJ, Mantegazza R, Meriggioli MN, Quan J, Wolfe GI; Task Force on MG Study Design of the Medical Scientific Advisory Board of the Myasthenia Gravis Foundation of America. Recommendations for myasthenia gravis clinical trials. Muscle Nerve. 2012 Jun;45(6):909-17. doi: 10.1002/mus.23330. PMID 22581550
- [Background] Troha Gergeli A, Neubauer D, Golli T, Butenko T, Loboda T, Maver A, Osredkar D. Prevalence and genetic subtypes of congenital myasthenic syndromes in the pediatric population of Slovenia. Eur J Paediatr Neurol. 2020 May;26:34-38. doi: 10.1016/j.ejpn.2020.02.002. Epub 2020 Feb 11. PMID 32070632
- [Background] Pane M, Coratti G, Brogna C, Mazzone ES, Mayhew A, Fanelli L, Messina S, D'Amico A, Catteruccia M, Scutifero M, Frosini S, Lanzillotta V, Colia G, Cavallaro F, Rolle E, De Sanctis R, Forcina N, Petillo R, Barp A, Gardani A, Pini A, Monaco G, D'Angelo MG, Zanin R, Vita GL, Bruno C, Mongini T, Ricci F, Pegoraro E, Bello L, Berardinelli A, Battini R, Sansone V, Albamonte E, Baranello G, Bertini E, Politano L, Sormani MP, Mercuri E. Upper limb function in Duchenne muscular dystrophy: 24 month longitudinal data. PLoS One. 2018 Jun 20;13(6):e0199223. doi: 10.1371/journal.pone.0199223. eCollection 2018. PMID 29924848
- [Background] Mayhew AG, Coratti G, Mazzone ES, Klingels K, James M, Pane M, Straub V, Goemans N, Mercuri E; Pul Working Group. Performance of Upper Limb module for Duchenne muscular dystrophy. Dev Med Child Neurol. 2020 May;62(5):633-639. doi: 10.1111/dmcn.14361. Epub 2019 Sep 19. PMID 31538331
- [Background] Pierzchlewicz K, Kepa I, Podogrodzki J, Kotulska K. Spinal Muscular Atrophy: The Use of Functional Motor Scales in the Era of Disease-Modifying Treatment. Child Neurol Open. 2021 Apr 27;8:2329048X211008725. doi: 10.1177/2329048X211008725. eCollection 2021 Jan-Dec. PMID 33997096
- [Background] Burns TM, Sadjadi R, Utsugisawa K, Gwathmey KG, Joshi A, Jones S, Bril V, Barnett C, Guptill JT, Sanders DB, Hobson-Webb L, Juel VC, Massey J, Gable KL, Silvestri NJ, Wolfe G, Cutter G, Nagane Y, Murai H, Masuda M, Farrugia ME, Carmichael C, Birnbaum S, Hogrel JY, Nafissi S, Fatehi F, Ou C, Liu W, Conaway M. International clinimetric evaluation of the MG-QOL15, resulting in slight revision and subsequent validation of the MG-QOL15r. Muscle Nerve. 2016 Dec;54(6):1015-1022. doi: 10.1002/mus.25198. Epub 2016 Nov 7. PMID 27220659
- [Background] Wolfe GI, Herbelin L, Nations SP, Foster B, Bryan WW, Barohn RJ. Myasthenia gravis activities of daily living profile. Neurology. 1999 Apr 22;52(7):1487-9. doi: 10.1212/wnl.52.7.1487. PMID 10227640
- [Background] Ousmen A, Touraine C, Deliu N, Cottone F, Bonnetain F, Efficace F, Bredart A, Mollevi C, Anota A. Distribution- and anchor-based methods to determine the minimally important difference on patient-reported outcome questionnaires in oncology: a structured review. Health Qual Life Outcomes. 2018 Dec 11;16(1):228. doi: 10.1186/s12955-018-1055-z. PMID 30537955
- [Background] Cornett KMD, Menezes MP, Bray P, Shy RR, Moroni I, Pagliano E, Pareyson D, Estilow T, Yum SW, Bhandari T, Muntoni F, Laura M, Reilly MM, Finkel RS, Eichinger KJ, Herrmann DN, Shy ME, Burns J; CMTPedS Study Group. Refining clinical trial inclusion criteria to optimize the standardized response mean of the CMTPedS. Ann Clin Transl Neurol. 2020 Sep;7(9):1713-1715. doi: 10.1002/acn3.51145. Epub 2020 Aug 6. PMID 32762141
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002093-N.html